CLINICAL TRIAL: NCT00925821
Title: Lenalidomide (Revlimid®), Adriamycin and Dexamethasone (RAD)as an Induction Therapy in Newly Diagnosed Multiple Myeloma Followed by a Risk-Defined Transplant Strategy and Lenalidomide Maintenance - A Multicenter Phase II Trial by Deutsche Studiengruppe Multiples Myeloma (DSMM XII)
Brief Title: Lenalidomide-Adriamycin-Dexamethasone (RAD) Induction Followed by Stem Cell Transplant in Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: ClinAssess GmbH (Industry); Celgene Corporation (Industry); Amgen (Industry); medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSMM XII
Record Dates: First submitted 2009-06-16; First posted 2009-06-22 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Multiple Myeloma
Keywords: Allogeneic stem cell transplantation; Lenalidomide; IMiD
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allogeneic stem cell transplant (Experimental): Second scheduled transplantation performed from an HLA-matched MRD or MUD after conditioning with treosulfan and fludarabine
  Interventions: Procedure: allogeneic stem cell transplant versus second autologous transplantation; Drug: RAD
- High-dose melphalan chemotherapy (Active Comparator): Second high-dose melphalan therapy followed by transplantation of peripheral blood stem cells
  Interventions: Procedure: allogeneic stem cell transplant versus second autologous transplantation; Drug: RAD

INTERVENTIONS:
Procedure: allogeneic stem cell transplant versus second autologous transplantation — Transplantation of stem cells from a MRD or MUD, respectively after dose-reduced conditioning versus autologous stem cell graft after preparation with melphalan 200 mg/m²
Drug: RAD — After enrollment, patients are to receive four cycles of RAD induction treatment: a combination of lenalidomide (Revlimid), adriamycin, and dexamethasone.

SUMMARY:
Subjects up to the age of 65 years with newly diagnosed multiple myeloma requiring treatment are eligible. Minimal pretreatment (2 cycles of chemotherapy; local irradiation; surgery) is permitted. After enrollment, patients are to receive four cycles of RAD induction treatment: a combination of lenalidomide (Revlimid), adriamycin, and dexamethasone. If at least a minimal response is achieved to RAD, they will undergo chemomobilization (cyclophosphamide, etoposide) of peripheral blood stem cells and one uniform cycle of high-dose melphalan chemotherapy followed by a first stem cell transplant. If any of the high-risk features (such as elevated beta 2-microglobulin, adverse cytogenetic factors, elevated LDH, Ig A isotype) were present at diagnosis, patients will be allocated to a consolidative allogeneic transplant following dose-reduced conditioning. If no appropriate donor is available, the patient does not consent or lacks of high-risk features a second autograft following high-dose melphalan will be delivered. All patients will proceed to lenalidomide maintenance (one year) following hematopoietic reconstitution.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Newly diagnosed multiple myeloma
* Maximum of one prior systemic therapy (2 cycles)
* Presence of CRAB criteria
* Measurable disease parameters
* Left ventricular ejection fraction at least 55%
* DLCO of at least 60%
* Adequate bone marrow function
* Use of adequate contraception for female subjects with childbearing potential and all male subjects
* Eligible for autologous and allogeneic stem cell transplantation
* Bone marrow baseline sample evaluable for interphase cytogenetics

Exclusion Criteria:

* Any serious medical conditions preventing the subject from written informed consent
* Progressive disease (PD) to any initial treatment
* Pregnant or lactating females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data
* Use of any other experimental drug or therapy within 28 days of baseline
* Preexisting neuropathy of ≥ grade 2 severity
* Known hypersensitivity to thalidomide
* Any prior use of lenalidomide
* Positive for HIV or infectious hepatitis, type A, B or C after serologic testing
* Serum creatinine despite induction therapy ≥ 2.0 mg/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2009-06

PRIMARY OUTCOMES:
Response rate to RAD induction and transplant (stringent CR, CR, very good PR) | 9 months from start of treatment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 9 months from start of treatment
Incidence and relationship of severe adverse events | 1 year from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ralf C Bargou, MD, Principal Investigator — Wuerzburg University Hospital, Dept. of Internal Medicine II
Locations (12):
- Germany (12):
  - Charité University Hospital - Virchow Klinikum, Berlin
  - Dresden University Hospital, Dresden
  - Erlangen University Hospital, Erlangen
  - Freiburg University Hospital, Freiburg im Breisgau
  - Jena University Hospital, Jena
  - Kiel University Hospital, Kiel
  - Munich Grosshadern University Hospital, Munich
  - University Hospital of Munich Technical University, Munich
  - Klinikum Nuremberg, Nuremberg
  - Regensburg University Hospital, Regensburg
  - Rostock University Hospital, Rostock
  - Ulm University Hospital, Ulm

REFERENCES:
- See also: Website of the German Lymphoma Competence Net — http://www.lymphome.de/Gruppen/MMSG/index.jsp